CLINICAL TRIAL: NCT05285527
Title: MiSight 1 Day Safety Post-Approval Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAS002
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MiSight 1 Day (Experimental): MiSight 1 Day
  Interventions: Device: MiSight 1 Day

INTERVENTIONS:
Device: MiSight 1 Day — Subjects will wear MiSight 1 day lenses for three years.

SUMMARY:
The purpose of this post-approval study is to confirm the safety of daily disposable soft contact lens wear among the intended patient population for the MiSight 1 Day lens in the US.

DETAILED DESCRIPTION:
This prospective post-approval study of safety in a US study population is to confirm the safety of MiSight 1 day lenses. Consecutive subjects receiving the MiSight 1 Day lens, who meet the inclusion criteria, will be prospectively offered to participate in the study. Additionally, safety data from the MiSight 1 Day Post-Approval Study for Effectiveness and Visual Symptoms (PAS001) will be used to supplement this safety study.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 8 and 12 years of age inclusive at the time of enrollment.
2. Manifest Refraction - Spherical Equivalent Refractive Error (SERE) at baseline between -0.50 D and -7.00 D inclusive (at the corneal plane).
3. Best-corrected visual acuity by manifest refraction of at least 20/25 bilaterally
4. Free of ocular disease or abnormalities (including any corneal scar)
5. The parent/guardian must be capable of comprehending the nature of the study and consent to the use and release of their child's de-identified health care encounter data to be used for purposes of this study. Assent will be obtained from the child in a manner specified by the IRB.
6. Parent/Guardian must sign the Release of Medical Records associated with the outcomes of interest identified from claims data.
7. Interested in wearing contact lenses for approximately 10 hours per day and 6 days per week.
8. Possesses, or obtains prior to dispensing, wearable and visually functional (20/40 or better) eyeglasses.

Exclusion Criteria:

1. Acute and subacute inflammation or infection of the anterior chamber of the eye.
2. Any eye disease, injury, or abnormality that affects the cornea, conjunctiva, or eyelids.
3. Severe insufficiency of lacrimal secretion (dry eyes).
4. Corneal hypoesthesia (reduced corneal sensitivity), if not aphakic.
5. Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
6. Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.
7. Any active corneal infection (bacterial, fungal, or viral).
8. If eyes are red or irritated.
9. The patient is unable to follow lens handling and wear regimen or unable to obtain assistance to do so.
10. In addition to the labeling contraindications, children who are under medication that would interfere with contact lens wear, or who are using any pharmaceuticals for control of myopia will not be included in the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Microbial Keratitis (MK) | 3 years
  Incidence of Microbial Keratitis (MK) ≥ 1 mm

SECONDARY OUTCOMES:
Incidence of peripheral infiltrative keratitis/non-infectious ulcers | 3 years
  Incidence of peripheral infiltrative keratitis/non-infectious ulcers ≤ 1 mm
Incidence of non-infectious infiltrative keratitis | 3 years
  Incidence of non-infectious infiltrative keratitis ≤ 1 mm
Incidence of loss of best-corrected visual acuity | 3 years
  Incidence of loss of best-corrected visual acuity ≥ 2 lines for any adjudicated adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: William Gleason, OD, Principal Investigator — Foresight Regulatory Strategies
Locations (50):
- United States (47):
  - Experts on Sight LLC., Gilbert, Arizona
  - Centerton Family Eyecare, Centerton, Arkansas
  - University of California, Berkeley University Eye Center, Berkeley, California
  - Golden Vision Cupertino Optometry, Cupertino, California
  - Boghossian Vision, Danville, California
  - Iron Horse Optometric Group, Dublin, California
  - Capitol Eye Care Center Optometry, Fremont, California
  - Irvine Eye Physicians and Surgeons Inc, Irvine, California
  - Elsa Pao OD, Inc, Oakland, California
  - Perfect Pair Optometry, San Jose, California
  - Almaden Family Optometric Center, San Jose, California
  - Children's Eye Physicians, Centennial, Colorado
  - Eye Physicians & Surgeons, PC, Milford, Connecticut
  - Planet Vision Eyecare, Lake Worth, Florida
  - Marino Eye Care, Miami, Florida
  - Vision Source Oviedo, INC, Oviedo, Florida
  - Dau Family Eye Care, Saint Johns, Florida
  - Gulf Coast Eye Center, Sarasota, Florida
  - Weston Contact Lens Institute LLC, Weston, Florida
  - Lurie Childrens, Chicago, Illinois
  - Lyons Family Eye Care P.C., Chicago, Illinois
  - Darien Eye Specialists, Darien, Illinois
  - Carillon Vision Care, Glenview, Illinois
  - Little Eyes Pediatric Eye Care, Carmel, Indiana
  - All Eyes on Rockville, Rockville, Maryland
  - Wellesley Vision Group at Optical Design, Wellesley, Massachusetts
  - Missouri Eye Consultants - California, California, Missouri
  - Center for Vision and Learning, Des Peres, Missouri
  - Advocare Pediatric Eye Physicians, Morristown, New Jersey
  - Bronx Eye Associates, The Bronx, New York
  - Clarity Vision, Apex, North Carolina
  - Cary Family Eye Care, Cary, North Carolina
  - Chagrin Valley Optometrists, Inc., Chagrin Falls, Ohio
  - Pickerington Eye Care, Pickerington, Ohio
  - Nittany Eye Associates, LLC, State College, Pennsylvania
  - Texas State Optical, Beaumont, Texas
  - Bellaire Family Eye Care, Bellaire, Texas
  - Drs. McIntyre, Garza, Avila and Jurica, Optometrists, Corpus Christi, Texas
  - Clarkson EyeCare KIDS, Frisco, Texas
  - Lone Star Vision Center, Plano, Texas
  - Stone Oak Vision Source, San Antonio, Texas
  - Child & Family Eye Care Center, Pleasant Grove, Utah
  - Broadway Eye Clinic, Salt Lake City, Utah
  - Invision Eye Health, Sandy City, Utah
  - Colonial Eye Care, Williamsburg, Virginia
  - Redmond Eye Clinic, Redmond, Washington
  - Spectrum Optical, PLLC, Morgantown, West Virginia
- Canada (3):
  - Dr. Kit Guan & Associates, Markham, Ontario
  - Abbey Eye Care, Oakville, Ontario
  - Optometry Professional Corporation, Toronto, Ontario